CLINICAL TRIAL: NCT02529319
Title: Efficacy of Delayed Enhancement MRI-Guided Ablation vs Conventional Catheter Ablation of Atrial Fibrillation: The DECAAF II Study
Brief Title: Efficacy of Delayed Enhancement MRI-Guided Ablation vs Conventional Catheter Ablation of Atrial Fibrillation
Acronym: DECAAFII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Collaborators: Tulane University (Other)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB_00076945
Record Dates: First submitted 2015-08-11; First posted 2015-08-20 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation; Fibrosis
Keywords: atrial fibrillation; ablation
MeSH Terms: conditions — Atrial Fibrillation; Fibrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI-Guided Ablation (Experimental): Surgery
  Patients will undergo catheter ablation using DE-MRI as a guide for fibrosis imaging.
  Interventions: Procedure: MRI-Guided Ablation
- Conventional Ablation (Active Comparator): Surgery
  Patients will undergo conventional catheter ablation as described by the HRS guidelines.
  Interventions: Procedure: Conventional Ablation

INTERVENTIONS:
Procedure: MRI-Guided Ablation — Catheter ablation of AF will be guided by a DE-MRI of the patient's heart prior to the procedure.
  Arms: MRI-Guided Ablation
Procedure: Conventional Ablation — Catheter ablation of AF using pulmonary vein isolation (PVI) will be performed using the HRS guidelines.
  Arms: Conventional Ablation

SUMMARY:
This proposal is aiming at modifying and improving persistent AF management guidelines by evaluating targeting DE-MRI detected atrial fibrosis during AF ablation and its related effect on procedural outcome.

OBJECTIVES:

Primary Objective: To examine the efficacy of targeting atrial fibrosis tissue during an ablation procedure in treating persistent AF. Results from the DECAAF study show that one of the most important predictors of ablation outcome was the degree of ablation of the fibrotic tissue; the more fibrotic tissue that was overlapped with scar during ablation, the better the outcome. These results were the impetus for the primary outcome of DECAAF II. Patients will be randomized to receive conventional pulmonary vein isolation (PVI) ablation or PVI + fibrosis-guided ablation. The investigators will follow patients longitudinally to assess the primary outcome identified as recurrence of persistent atrial arrhythmias (AA) (atrial fibrillation, atrial flutter or atrial tachycardia as defined by recent guidelines [2]). The investigators hypothesize that patients receiving fibrosis-guided ablation in addition to conventional PVI ablation will have fewer AA recurrences than those who receive PVI ablation alone.

The investigators will also examine the efficacy of the fibrosis-guided ablation intervention on a number of secondary or exploratory outcomes including the individual components of the primary outcome (atrial fibrillation, atrial flutter and atrial tachycardia), symptomatic atrial arrhythmia, AF cycle length/regularity/termination, cardiovascular (CV)-related hospitalization, CV-related mortality, quality of life measurements (University of Toronto Atrial Fibrillation Severity Scale (AFSS), and AF burden.

The safety of the two interventions will be evaluated by evaluating peri-procedural complications including stroke, peripheral vascular stenosis, bleeding, esophageal injury, cardiac perforation, heart failure, and death.

DETAILED DESCRIPTION:
BACKGROUND AND INTRODUCTION:

Atrial fibrillation (AF) is the most common cardiac arrhythmia affecting millions of people in the US and around the world. Treating AF continues to be a challenge. Over the last 15 years, catheter based AF ablation procedure has been widely adopted. Approximately 50% of patients treated with catheter ablation present with a persistent type of the arrhythmia. Unfortunately, ablation results in this population have been dismal, not only because of low success rates in suppressing arrhythmias, but also from a healthcare cost point of view. In fact, the long-term success of such a procedure has been reported to be as low as 20%, and patients may need more than two ablation procedures to achieve temporary arrhythmia suppression. The cost of AF ablation among Medicare patients followed for a year after ablation was found to be US$16,049 ± 12,536 if ablation was successful versus US$19,997 ± 13,958 for failed ablation. A major issue contributing to the low success of catheter ablation is the lack of a protocol to appropriately select patients that would respond to this treatment. Currently, cardiologists base their decision to ablate persistent AF on various comorbidities, a concept that has not been proven successful. With the introduction of AF ablation as a first line therapy option in the recent guidelines, a better and more accurate selection protocol is urgently needed. There is a strong association between AF and atrial tissue fibrosis. Recently, a novel DE-MRI (Delayed-Enhancement MRI) based imaging modality has been demonstrated to reveal the degree of fibrotic atrial tissue in patients suffering from AF. When applied in various studies, including a multicenter study, extent of fibrotic atrial changes was shown to be the strongest independent predictor of a successful treatment in patients undergoing ablation of AF. Moreover, in the multicenter observational study DE-MRI Determinant of Successful Radiofrequency Catheter Ablation of Atrial Fibrillation (DECAAF), the strongest independent predictor of successful outcome was the surface area of fibrosis covered by ablation lesions. In fact, the number of encircled pulmonary veins, the most common adopted approach to ablate AF today, did not predict catheter ablation success.

The use of non-invasive ambulatory electrocardiography (ECG) devices including 24-48 hour Holter monitors and 30-day cardiac event monitors have been widely used for the detection of cardiac rhythm abnormalities. The duration of time for rhythm evaluation is key to detect arrhythmias and conduction abnormalities, as number of arrhythmia diagnoses increases with increasing duration of monitoring. The longer duration of monitoring occurs at the expense of patient comfort and patient compliance. Previous FDA- approved devices for standard of care monitoring are limited in the duration of monitoring. At many institutions, it is standard of care to wear a 60-day cardiac event monitor for the detection and evaluation of cardiac arrhythmias in the post-ablation blanking period.

The percentage of asymptomatic recurrences of AF drastically increases after ablation. Thus, post-procedure devices are necessary for close monitoring and detection of asymptomatic AF in ablation patients. Compliance with the current cardiac event monitors may be low for many reasons. Electrode intolerance due to skin rashes, irritation and/or breakdown, and the unwillingness for continuous devices to be worn are some known areas of non-compliance.

A higher level of monitoring can be provided with use of new wireless ECG technologies, specifically, the FDA approved ECG Check mobile heart monitor designed by Cardiac Designs. This mobile heart monitor will enable patients to record their heart rhythm anytime and anywhere. The device will automatically analyze the ECG for symptomatic or asymptomatic arrhythmias for the duration of their life as long as it is compatible with their current "smart phone" or tablet computer. This is a patient-owned monitor.

The ECG Check is the first FDA-approved over-the-counter ECG monitor that is currently compatible with approved smart phones. This will allow patients to record, store, transfer and analyze single-channel ECG wirelessly through the ECG Check app and the ECG Check Web Center. The information will be uploaded to a protected server through Cardiac Designs.

DESIGN:

DECAAF II is a prospective, randomized, multicenter trial of patients with persistent AF and presence of atrial fibrosis. After consenting to participate in the study, the subject will undergo a DE-MRI scan to assess for extent of atrial fibrosis. Consented patients will be randomized to one of two study groups to receive conventional PVI ablation (Group 1) or PVI + fibrosis-guided ablation (Group 2). In Group 1, PVI ablation will be performed as recommended by the Heart Rhythm Society (HRS) consensus statement and physicians will be blinded to the pre-ablation MRI fibrosis results. In Group 2, physicians will receive the DE-MRI scan prior to the ablation procedure and will complete conventional PV isolation and will target left atrial fibrosis detected by MRI during the ablation procedure.

Once randomized, the follow-up period for each patient will extend for 18 months following the patient's ablation procedure or until a common administrative censoring date 12 months after the ablation procedure of the final randomized subject, whichever comes first. If a randomized patient fails to undergo ablation, the patient will be followed for 18 months from the patient's randomization date or until 12 months after the last patient is randomized, whichever comes first.

This is an event-driven trial, in which patient enrollment and follow-up will continue until approximately 517 randomized subjects experience the primary endpoint of AA recurrence. Under the assumptions described in the analysis section, it is anticipated that 888 subjects will be randomized, including 444 assigned to Group 1 and 444 assigned to Group 2. The actual number enrolled and the duration of the follow-up period will be adjusted as necessary to achieve the 517 required events.

STUDY PROCEDURES

Recruitment Clinical Center staff will approach all potentially eligible patients to participate in the study. The de-identified characteristics of those refusing to participate will be collected to ascertain if there is any selection bias that would limit applicability of the results.

Consent If the patient has met the eligibility criteria, the Clinical Center investigator or delegated study staff will approach the patient to explain the study and obtain informed consent from the subject to participate. The investigator or designated staff will provide an explanation of study procedures of the benefits and risks, and the costs and compensation involved with the study. Participants will be given sufficient time to read the consent form and the individual obtaining the informed consent will answer any questions posed by the participant.

Imaging Protocol All patients will undergo a DE-MRI within 30 days prior to the ablation procedure using the Marrek DE-MRI protocol (MRI sequence and Image processing software). The purpose of the initial MRI is to quantify the degree of atrial structural remodeling or fibrosis prior to the ablation. If a patient has a heart rate ≥ 90 beats per minute, they will be pre-medicated with a beta blocker prior to the MRI in order to obtain optimal images. Images will be sent to Marrek Inc., (Salt Lake City, UT) and will be reviewed for quality by trained technicians using a standard protocol. Images that do not meet quality standards will not be further processed. The site physician may opt to repeat the MRI scan and re-submit it for evaluation. If the image meets quality standards and can be processed, then Marrek will verify that the subject has some proportion of atrial fibrosis (not limited to advanced stage fibrosis). Utah Stages 1-4 will be used to classify patients based on percent fibrosis. Subjects for whom images are successfully evaluated and scored for fibrosis will be randomized. Following ablation, DE-MRIs will be obtained at the 90 day follow up to detect and quantify ablation-related scar formation.

Randomization After images have been processed and scored for fibrosis, the Data Coordinating Center (DCC) staff will complete randomization procedures using a web-based randomization service. Randomization will be stratified by Clinical Center and by Utah Stage (with two Utah stage strata defined by Utah stages I - II and Utah stages III - IV). For subjects who are randomized to the fibrosis-guided ablation arm (Group 2), DCC will make the processed images available to the investigator at the Clinical Center for use during the ablation procedures. Processed fibrosis images of subjects who are randomized to the PVI ablation group (Group 1) will not be made available to clinicians or site staff. All images will be retained at the Marrek site for storage and later analysis. Clinical investigators will schedule the ablation procedures to occur within approximately 30 days after imaging has been completed.

The study outcome is formally defined by at least two consecutive, valid ECG tracings indicating an atrial arrhythmia (AA) (atrial fibrillation, atrial flutter or atrial tachycardia). Both tracings must be completed after the 90-day blanking period. The two consecutive tracings demonstrating an atrial arrhythmia must be recorded between 6 hours and 7 days of each other. If an ECG Check tracing demonstrates a non-self-terminating bout of an atrial arrhythmia (AA), the DCC systems will send a notification to the Clinical Center indicating that an atrial arrhythmia has been observed. If a second, consecutive ECG Check reading also demonstrates an atrial arrhythmia 6 hours or up to 7 days after the first recording, the DCC system will again notify the Clinical Center. In cases where a 12-lead ECG, obtained for clinical or other reasons, first demonstrates an atrial arrhythmia, a subsequent, consecutive, valid ECG reading will also be confirmatory of having met the study outcome. The 12-lead ECG data will be transmitted to the DCC for inclusion in the study database. This ECG will not be transmitted to the central location for review; rather any 12-lead obtained in association with a study outcome will be read by an independent expert to verify the presence of AA. This expert will be blinded to study arm. In the possible scenario where a second ablation is performed after the 90-day blanking period, but there is no recurrence demonstrated by either ECG measure (12 lead or ECG Check), AA recurrence will be inferred and assigned to the date of the second ablation.

Devices utilized in this trial In this trial, 3 different U.S. Food and Drug Administration (FDA) approved devices will be utilized. The first is a hand-held ECG application that transmits the ECG. This device has been approved for the transmittal of ECG information. The second is a software application for viewing and post-processing of cardiovascular MRIs to obtain left atrial enhancement quantification and visualization on a 3D model, which has been previously approved for this indication. Finally, ablation catheters that are used for atrial fibrillation treatment are being used in their approved manner. Although this trial will be the first to use all 3 devices together, this use does not necessitate a new IDE as this composite utilization falls within current approvals for each device for their approved indications.

Study Endpoints The primary endpoint of the study is the recurrence of atrial arrhythmia post-ablation, defined as a non-self-terminating bout of atrial fibrillation, atrial flutter, or atrial tachycardia demonstrated by at least two consecutive, valid ECG tracings occurring within 6 hours up to a maximum of 7 days of each other after the 90-day post-ablation blanking period. The primary endpoint will be determined from tracings from the ECG Check mobile device or a clinically obtained 12-lead ECG indicating persistent atrial arrhythmia. The clinically obtained 12-lead ECG option will be used if the subject is unwilling or unable to continue to use the ECG check device. It is difficult to anticipate whether the subject population will have technical difficulty or accessibility issues using the smart phone and tablet devices on a daily basis; the 12-lead ECG option is geared to offer an option for those unable to continue to use the device. If a subject undergoes a second ablation procedure during the study period (after the 90-day blanking period) but does not have a documented atrial arrhythmia by the methods described previously, the ablation will also constitute a study endpoint. Ablations occurring within the 90 day blanking period will not be counted as an outcome.

Project Enrollment and Follow-up Timeline: This will be a 3-year study with approximately 9 months allotted for developing materials, Institutional Review Board (IRB) approvals, startup activities, and rolling patient enrollment, approximately 12 months for follow-up after the last patient is randomized, and 6 months for close-out activities and manuscript preparation. Our success with DECAAF and the basic inclusion criteria highlight the feasibility of this project to be completed within 3 years. In addition, many of these Clinical Centers participated in DECAAF and presented successful recruitment.

STATISTICAL ANALYSIS AND POWER

Analysis Populations Randomized Study Population The randomized study population consists of all randomized patients, irrespective of whether the patient receives an ablation procedure or remains in the trial at the close of the blanking period.

Safety Population. The safety population consists of all randomized patients who receive an ablation procedure.

Modified Intent-to-Treat Population. The modified intent-to-treat population consists of all randomized patients who remain in follow-up at the close of the 90-day blanking period irrespective of whether or not the ablation was actually performed.

Unless indicated otherwise, all statistical analyses of efficacy outcomes will be performed in the modified intent-to-treat population and all analyses of safety outcomes will be carried out in the safety population.

Descriptive Analyses of Baseline Characteristics Descriptive summaries of baseline clinical and demographic characteristics will be provided by randomized treatment assignment for a) the randomized study population, b) the safety population, and c) the modified intent-to-treat population. Baseline characteristics will also be summarized by randomized group in the modified intent-to-treat population for each region (North America, Europe, Asia) and for each clinical center. In the event that substantial imbalances in particular factors between the randomized treatment groups are detected, sensitivity analyses will be performed after adding these factors as covariates to the Cox regression analyses described in the Primary Analysis section below.

Primary Analysis of Atrial Arrhythmia Recurrence The primary efficacy analysis will be performed in the modified intent-to-treat population using a stratified log-rank test to compare the time to the first atrial arrhythmia recurrence after the blanking period between the randomized treatment groups. The log rank test will be stratified by Utah Stage (separate strata for Utah stages I, II, III, and IV) and region (US/Asia/Canada and Europe). Follow-up will be censored at loss-to-follow-up or death. The primary analysis will be performed with a 2-sided significance level (alpha) of 0.05.

An associated Cox proportional hazard regression analysis with the same stratification factors will be performed to estimate the hazard ratio between the fibrosis guided ablation and conventional ablation groups with its 95% confidence interval. The possibility that the hazard ratio for treatment assignment varies over the follow-up period (non-proportional hazards) will be investigated by smoothed Schoenfeld residual plots and by performing time-dependent Cox regressions including interaction terms between treatment assignment and follow-up time [S1, S2]. Cumulative incidence curves for the first atrial arrhythmia recurrence and for death will be constructed by randomized group using a competing risk framework [S3, S4].

Components of Atrial Arrhythmia Recurrence The frequencies and proportions of patients experiencing each of three components of the primary atrial arrhythmia outcome - 1) atrial fibrillation, 2) atrial flutter, and 3) atrial tachycardia - will be tabulated by treatment group. As in the primary analysis, only events occurring after the end of the blanking period will be counted in these analyses. Cox regression analyses in which the baseline hazard function is stratified by Utah stage and region will be used to obtain estimates of cause-specific hazard ratios and associated 95% confidence intervals to compare the three components of the primary outcome between the randomized treatment groups. Cumulative incidence curves will be constructed for each of the three components and death under a competing risk framework [S3, S4]. The same analyses will also be performed for symptomatic atrial arrhythmia and for symptomatic atrial arrhythmia requiring treatment. Because the analyses of the components of the primary endpoint are explanatory, no adjustment for multiple comparisons will be performed.

Subgroup Analyses of Atrial Arrhythmia Recurrence Stratified log-rank tests and Cox-regressions similar to those described for the primary analysis will be used to compare the fibrosis guided ablation and conventional interventions in subgroups defined by baseline fibrosis ≤ or > 20%. The log-rank test and Cox regression in the fibrosis ≤ 20% subgroup will be stratified by Utah Stages I and II, while the analyses of the fibrosis > 20% subgroup will be stratified by Utah Stages III and IV. These analyses will be repeated for the three components of the primary outcome.

Within-Treatment Group Analyses of Atrial Arrhythmia Recurrence Cumulative incidence curves for the first Atrial Arrhythmia recurrence and for death will be constructed by randomized group separately for each of the four Utah stages in order to estimate the proportions of subjects reaching these events by 1 year and by 18 months within each Utah stage. Separate Cox regression models using cubic splines for percent fibrosis will be used to relate the hazard for Atrial Arrhythmia recurrence to the pre-ablation percent fibrosis within each randomized group. Similar Cox regressions with cubic splines will be performed within each randomized group to relate the hazard for Atrial Arrhythmia recurrence to the percentage of fibrosis which is covered by the ablation procedure.

Main Secondary Efficacy Outcome Quality of life as measured by the Toronto Score will be treated as the main secondary efficacy outcome. The main secondary analyses will estimate the effect of the treatment on the mean Toronto scores at months 3, 12, and 18 under a mixed effects model in which the baseline Toronto score, visit month (treated as a categorical variable) and the interaction between treatment and visit month are included as fixed effects. An unstructured covariance model will be used to account for serial correlation in the Toronto scores across the follow-up visits. The main contrast for testing the effect of the treatment will compare the adjusted mean Toronto scores at month12 between the guided ablation and usual care groups. A secondary contrast will compare the adjusted mean Toronto scores at months 3 and 12 between the guided ablation and usual care groups.

Additional Efficacy Outcomes Stratified log-rank tests and associated Cox-regressions will also be used to compare initial occurrences of a) a composite outcome including AA recurrence and prescription of an anti-arrhythmic medication, b) stroke, c) cardiovascular hospitalization, d) a repeat ablation, and e) AA recurrence following repeat ablation between the randomized treatment groups. The analysis of repeat ablations will evaluate the time from the end of the blanking period to the first ablation performed after the close of the blanking period. The analysis of AA recurrence following repeat ablation will evaluate the time from the end of the blanking period to the first AA recurrence following the first repeat ablation. If the patient has an AA recurrence after the blanking period but does not have a repeat ablation, the outcome for this analysis will be defined as the initial AA recurrence after the blanking period.

Mixed effects analyses similar to those described for the Toronto scores will be performed to compare the physical and mental composite scores from the San Francisco-36 (SF-36) between the randomized group at months 3, 12 and 18, with primary emphasis given to the month-12 comparison.

The proportions of positive responses to the 5 questions asked every other week pertaining to chest pain, shortness of breath, heart racing, dizziness, and syncope will displayed graphically along with associated exact binomial 95% confidence intervals by follow-up week and treatment group. The mean proportions of positive responses over the full follow-up period will be compared between the targeted ablation group and the usual care group using generalized estimating equations with a working identity covariance matrix, with covariate adjustment for the baseline responses [S5]. The Huber sandwich estimator will be used to compute robust standard errors for statistical inferences.

AA burden will be estimated for each month of follow-up for each subject as a time-weighted average of the proportion of ECG Check readings during that follow-up month which indicate the presence of atrial arrhythmia. Generalized estimating equations with stabilized inverse probability of censoring weights to account for early loss-to-follow-up will be used to compare these proportions between the randomized treatment groups.

Safety Outcomes The primary safety composite outcome is defined by occurrence of one or more of the following events during the 1 week period following the ablation procedure: 1) stroke, 2) peripheral vascular stenosis, 3) bleeding, 4) heart failure and 5) death. Additional safety outcomes include each of the individual components of the primary safety composite as well as the occurrence of 6) cardiac perforation, or 7) esophageal injury within 1 week of the ablation procedure. The primary safety composite and the other safety outcomes will be compared between the randomized treatment groups among patients in the safety population using Fisher exact tests. The distributions of the duration of the ablation procedure and fluoroscopy time will also be summarized by randomized group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with persistent Atrial Fibrillation (AF) defined as 7 days or more of AF as evidence by rhythm strips or written documentation; AND
2. Undergoing first AF ablation as per recent HRS consensus document; AND
3. Age ≥ 18 years

Exclusion Criteria:

1. Previous left atrial ablation or any type of valvular surgery; OR
2. Contraindication for DE-MRI with a full dose contrast agent; OR
3. Contraindication to beta blockers, if necessary, for DE-MRI; OR
4. Women currently pregnant; OR
5. Mental or physical inability to take part in the study; OR
6. Inability to be placed in MRI due to body mass or body habitus; OR
7. Known terminally ill patients; OR
8. Subjects without daily access to a smart phone or tablet compatible with the ECG. Check application ability to upload ECG tracings for the entire follow up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 843 (Actual)
Dates: Start 2016-07; Primary Completion 2021-02-08 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
AF Recurrence | 18 months
  recurrence of 30 seconds of any atrial arrythmia as evidenced by a 45 second ECG strip.

CONTACTS AND LOCATIONS:
Overall Officials: Nassir Marrouche, MD, FHRS, Principal Investigator — Associate Professor
Locations (1):
- CARMA Center, University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Marrouche NF, Wazni O, McGann C, Greene T, Dean JM, Dagher L, Kholmovski E, Mansour M, Marchlinski F, Wilber D, Hindricks G, Mahnkopf C, Wells D, Jais P, Sanders P, Brachmann J, Bax JJ, Morrison-de Boer L, Deneke T, Calkins H, Sohns C, Akoum N; DECAAF II Investigators. Effect of MRI-Guided Fibrosis Ablation vs Conventional Catheter Ablation on Atrial Arrhythmia Recurrence in Patients With Persistent Atrial Fibrillation: The DECAAF II Randomized Clinical Trial. JAMA. 2022 Jun 21;327(23):2296-2305. doi: 10.1001/jama.2022.8831. PMID 35727277
- [Derived] Marrouche NF, Greene T, Dean JM, Kholmovski EG, Boer LM, Mansour M, Calkins H, Marchlinski F, Wilber D, Hindricks G, Mahnkopf C, Jais P, Sanders P, Brachmann J, Bax J, Dagher L, Wazni O, Akoum N; DECAAF II Investigators. Efficacy of LGE-MRI-guided fibrosis ablation versus conventional catheter ablation of atrial fibrillation: The DECAAF II trial: Study design. J Cardiovasc Electrophysiol. 2021 Apr;32(4):916-924. doi: 10.1111/jce.14957. Epub 2021 Mar 2. PMID 33600025